CLINICAL TRIAL: NCT06600308
Title: Walking ANalysis Interest in Persons wiTh facioscapulohumEral Muscular Dystrophies
Acronym: WANTED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HADOUIRI AOI 2022
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Facioscapulohumeral Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient (Experimental)
  Interventions: Other: Walk tests; Other: ecological (real-life) assessment of walking ability

INTERVENTIONS:
Other: Walk tests — Performance of the following walking tests using inertial measurement units: TUG; 10 m test at a comfortable and fast speed and TM6 (according to the recommendations of the American Thoracic Society).
  At the end of each walking test, measurement of the difficulty of exertion using the Borg scale.
Other: ecological (real-life) assessment of walking ability — Delivery of an actimeter, inertial units and logbook for ecological assessment (in real life) of walking ability for 7 days

SUMMARY:
Facioscapulohumeral muscular dystrophy (FSH) is one of the most common genetic myopathies in adults. It is characterised by progressive asymmetric muscular atrophy affecting the skeletal muscles of the face, upper limbs and then lower limbs, causing problems with walking, which is one of the most frequent complaints of these patients. In fact, 20% of people with FSH require a wheelchair from the age of 60. To date, scientific research into FSH has focused mainly on the molecular level, enabling potential therapeutic targets to be identified. Trials of gene therapies and other drug therapies are gradually emerging, with the aim of having a positive impact on these people's functional abilities, particularly walking difficulties. However, few studies have looked at the functional impact of FSH on these people, and in particular at the specific analysis of their walking ability In France, the functional assessment of FSH is carried out using a clinical reference scale called the Motor Function Measurement (MFM), the D1 sub-score of which studies items relating to standing and transfers. However, this scale does not objectively and specifically study gait disorders, and its application requires a great deal of time (at least 30 minutes) and specific training leading to certification, limiting its use in practice almost exclusively to centres of expertise and reference for neuromuscular diseases. The NeuroMuscular Score-D1 (NM-score D1), linked to the MFM D1 sub-score, is the only French scale validated in the literature for assessing the severity of gait disorders in FSH, but it is very little used in current practice because it is little known and only descriptive.

Certain functional tests of walking ability (so-called "short-duration" tests such as the 10-metre test at comfortable and fast speeds, the Time Up and Go test [TUG], and so-called "long-duration" tests such as the 6-minute test [TM6]) exist and are much simpler to use in clinical practice, do not require certification and can be carried out in a shorter time. However, to date there is no consensus on the use of these walking tests in FSH. Furthermore, their ecological capabilities (i.e. their ability to reflect what happens in real life) are not really known. In this sense, technological developments in quantified gait analysis (QGA) could help to assess locomotion disorders (of neurological, muscular or joint origin, etc.) more effectively and objectively. A more consensual use of gait tests in FSH with the use of innovative connected tools that are accessible (e.g. use of inertial units to measure spatio-temporal gait parameters during gait tests) in clinical routine would make it possible to obtain new gait analysis data to explore gait disorders more specifically and in a simple, rapid and objective manner, and thus improve and optimise the day-to-day monitoring of these patients by a large proportion of healthcare professionals.

The aim of the WANTED project is therefore to assess the value of quick and easy walking tests as part of the functional evaluation of patients with FSH by studying the correlation between the data obtained with these walking tests and that obtained with the MFM, the reference method, and also with data obtained in real-life conditions (e.g. physical activity time via actimetry).

ELIGIBILITY:
Inclusion Criteria:

Patient :

* Adult ;
* Having given written consent;
* With an established molecular genetic diagnosis of FSH;
* Able to understand the instructions for carrying out the various tests;
* Able to walk for at least 6 minutes, even intermittently;

Exclusion Criteria:

Patient :

* Not affiliated to or not benefiting from a social security scheme;
* With one or more cardiorespiratory contraindications to a 6-minute test;
* With another neuro-orthopaedic history (other than FSH) that could significantly compromise walking ability;
* With cognitive problems preventing them from performing standardised tasks;
* Under legal protection (curatorship, guardianship).
* Who are subject to a legal protection measure;
* Pregnant, parturient or breast-feeding woman;
* Unable to benefit from longitudinal follow-up (D15 and M6).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Average walking speed during TM6 | Through study completion, on average of 30 month

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France